CLINICAL TRIAL: NCT05185986
Title: Comparison the Home-based Pilates Exercises and the Combination of Home-based Pilates Exercises With Home-based Cognitive Rehabilitation Exercises on Executive Functions and Anxiety in Multiple Sclerosis Patients.
Brief Title: Investigating the Home-based RCTs of Pilates Exercises and Cognitive Rehabilitation Exercises for Executive Functions and Anxiety in MS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arak University of Medical Sciences (Other)
Collaborators: Pardis Specialized Wellness Institute (Other)
Responsible Party: Principal Investigator, Amir Hossein Kazemi, MSc. University of Arak, Arak University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 6436
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Executive Functions; Anxiety; Pilates; Cognitive Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator was blinded to participant allocation, and the analyses were performed blinded to the group. Participants' individual identification numbers assigned at baseline were used during the course of the trial. Identifying information were removed, such that no participant could be identified in the working dataset through one, or a combination of different variables.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home based Pilates exercises (Experimental): This group will perform two weekly sessions of Pilates for eight weeks, completed with at least 48-hours between sessions, in their own home, supported by a DVD developed and previously implemented and evaluated by the lead researcher in a feasibility trial among people with Multiple Sclerosis. Each Pilates session will last approximately one hour and is comprised of seven Pilates warm-up exercises and fourteen mat-based beginner's level exercise. Four repetitions of each Pilates movement will be performed during sessions in the first two weeks, with intensity being self-regulated by the participant based on level of physical condition. Repetitions will gradually progress at biweekly intervals, resulting in ten repetitions being performed for the final two weeks of the trial (Weeks 7 and 8). Six post-training stretches will be maintained for a minimum of thirty seconds.
  Interventions: Behavioral: Home-Based Pilates exercise
- Combination of Home-based Pilates exercises and Home-based Cognitive Rehabilitation exercises (Experimental): In addition to performing home-based Pilates exercises described in arm 1, this group will also perform home-based cognitive rehabilitation exercises for 8 weeks and 3 sessions per week. The interval between each session is at least 48 hours and each session will take between 30 to 45 minutes. Cognitive rehabilitation exercises are in pen and paper and each session includes two exercises in the areas of planning, cognitive organization, cognitive flexibility and working memory. All exercises will be explained to the subjects by a cognitive rehabilitation specialist, and in addition, explanations of all the exercises in each session will be available for participants in the separate voices. During the intervention period, in addition to the Pilates specialist, the cognitive rehabilitation specialist contacts the group 2 participants on a weekly basis and monitors their rehabilitation exercises.
  Interventions: Behavioral: Home-Based Pilates exercise; Other: Home-based Cognitive Rehabilitation
- Waiting list group (Other): This group is the waiting list group and acts as a control group and will be instructed to maintain their preintervention physical and cognitive activity levels during the intervention. After 8 weeks of intervention, Pilates exercises and cognitive rehabilitation exercises will be provided to the participants of this group for their own use.
  Interventions: Other: waiting list group

INTERVENTIONS:
Behavioral: Home-Based Pilates exercise — The Home-based Pilates is the two Pilates classes at home, twice weekly, for a period of eight weeks.
  Arms: Combination of Home-based Pilates exercises and Home-based Cognitive Rehabilitation exercises; Home based Pilates exercises
Other: Home-based Cognitive Rehabilitation — Home-based Cognitive Rehabilitation is the 3 sessions per week and 8 weeks of cognitive rehabilitation exercises at home. Each session consists of two Pen and paper exercises. Exercises are active in the areas of planning, cognitive organization, cognitive flexibility and working memory. Each session will take 30 to 45 minutes.
  Arms: Combination of Home-based Pilates exercises and Home-based Cognitive Rehabilitation exercises
Other: waiting list group — This group act as the control group and will maintain their physical and cognitive activities as the preintervention. Following the 8 weeks of intervention the home-based pilates and cognitive rehabilitation exercises will be provided to them for their own use.
  Arms: Waiting list group

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of home-based Pilates exercises and the combination of home-based Pilates exercises with home-based cognitive rehabilitation exercises, also to compare the effects of these two home-based interventions on executive functions and anxiety in MS patients. 51 MS patients of Isfahan MS society will be considered as sample and will be divided randomly into three groups of 17 participants. The first group is home-based Pilates exercises group, the second group is a combination of home-based Pilates exercises and home-based cognitive rehabilitation exercises and the third group is the waiting list group that is considered as the control group. Patients' scores on executive functions and anxiety will be assessed before and after 8 weeks of intervention.

DETAILED DESCRIPTION:
Since the onset of pandemic conditions in 2020 and the increase of lockdowns, almost all rehabilitation programs for MS patients in Iran were suspended, it is necessary to study the effects of home-based cognitive and physical interventions to improve executive functions and anxiety in MS patients. The present study will be conducted to investigate the effects of home-based Pilates exercises and the combination of home-based Pilates exercises with home-based cognitive rehabilitation as well as to compare the effects of these two interventions on executive functions and anxiety in MS patients. In this study, participants will be divided into two experimental groups and a control group. The research process and the reason for conducting the research will be explained to the candidates by lead researcher and the final participants will sign the research participation form. All 51 final participants will be identified by a code and their identity information will not be disclosed, and in order to avoid any bias, each code will be randomly divided into three groups randomly. Pre-test will be taken from all three groups before the intervention. Experiment group 1 will perform a home-based Pilates video training program for 8 weeks, two sessions a week at home, and will also pay attention to exercise-related tips for MS patients determined by specialists. At the same time, Experiment group 2 will be asked to perform home-based cognitive rehabilitation program for 8 weeks, 3 seasons a week at home, in addition to home-based Pilates exercises same as experimental group 1. Group 3 will also be on the waiting list as a control group and will not receive any interventions for 8 weeks. At the end of 8 week intervention, Pilates training packages and cognitive exercises will be provided to the control group for their own use. During the 8 weeks of the intervention, the Pilates instructor and the cognitive rehabilitation specialist will contact the subjects on a weekly basis and monitor their performance. Subjects will also be able to contact the researchers and express their questions and problems. Also, they will be able to hold online meetings with research facilitators for solving the problems and educating the exercises. During the 8 weeks of the intervention, if subjects have problems such as COVID-19 affection, coronary heart disease, muscle problems, relapse, and failure to perform more than 4 sessions of exercise, they will be excluded from the study by the lead researcher. In order to fully perform the exercises for people who do not perform up to 4 sessions of exercises, 2 weeks can be added to the intervention period, which will be applied by the lead researcher. After complete implementation of the intervention, post-test will be taken from all 3 groups and the results will be compared to the baseline and relative to each other.

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed Multiple Sclerosis
* EDSS score < 5
* Free from any other significant physical or psychiatric condition
* Have no previous Pilates experience

Exclusion Criteria:

* having cognitive or physical exercises at least from 3 months before intervention.
* Using psychiatric drugs or being under psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
change from baseline total number of cWMI | Baseline, week 8
  Computerized Working Memory Index (cWMI) The computerized figures width subscale of the Wechsler IQ scale, is used to measure working memory. Figures Width is the working memory subscale of the fourth edition of the Wechsler Intelligence Scale, which consists of two parts: Forward Figures Width and Inverted Figures Width and The sum of a person's scores in these two parts constitutes the total score of the person in this subscale.
change from baseline total time of cTOL | Baseline, week 8
  Computerized Tower Of London Task (cTOL) a computerized program in which patients are shown two pictures simultaneously of a goal board and a test board and are instructed to use the fewest possible moves to match the two boards. Each baseline and 8 week set of 12 problems consists of the same number of 2, 3, 4 or 5 move problems and has the same average difficulty level. Every problem could be repeated 3 times to be solved by participants. The dependent variables are the total number of task and the total time spent solving the problem (less time is better) and the delayed time or time to first move (less time is better).
change from baseline score of BAI | Baseline, week 8
  Beck Anxiety Inventory (BAI) Beck Anxiety Inventory (BAI) is a 21-item self-reported questionnaire which measures the existenceand severity of symptoms of anxiety. Each of the 21 items on BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and 26 - 63 as "Severe".

CONTACTS AND LOCATIONS:
Overall Officials: Tooraj Sepahvand, Phd., Study Director — University of Arak; Mohammad Ali Tabibi, Phd., Study Chair — Islamic Azad University of Khorasgan; Masoud Etemadifar, Phd., Study Chair — Isfahan University of Medical Sciences; Amir Hossein Kazemi, MS., Principal Investigator — University of Arak
Locations (1):
- MS society of Isfahan, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Participants' identities will not be shared. Each participant is identified by a code and the data obtained from the assessment of the participants by the research tools and the demographic data of the participants including age, education, marital status and EDSS score will be available via the email of the principal researcher.
Time Frame: starting march 2024
Access Criteria: Only for researchers who are studying on the related subjects. IPD sharing via principal investigator's email address will be available.

REFERENCES:
- See also: Multiple Sclerosis — https://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=multiple+sclerosis